CLINICAL TRIAL: NCT06714786
Title: Observational Study on Prevalence of Eating Behavior in Adult Patients With Diabetes Mellitus and/or Obesity, Listed or Already Undergoing Liver Transplantation
Brief Title: Observational Study of Eating Behavior in Patients With Diabetes Mellitus and Obesity Undergoing Liver Transplantation
Acronym: DCA-OLT-2020
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DCA-OLT-2020
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the presence of eating disorders, which consists of having an altered relationship with food, in patients on the list or already undergoing liver transplantation.

DETAILED DESCRIPTION:
The study involves the enrollment of at least 100 patients, currently followed for the treatment of severe organ failure, on the list or already undergoing liver transplantation and referred for a dietetic visit.

ELIGIBILITY:
Inclusion Criteria:

* signature of written informed consent to participate in the observational study, either by the participant or legal guardian

  * age > 18 years
  * diagnosis of type 2 diabetes mellitus and/or overweight or obesity, (BMI > 25)
  * be listed for OLT or have already been submitted to OLT

Exclusion Criteria:

* -previous diagnosis of psychiatric illness;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the enrollment of at least 100 patients, currently followed for the treatment of severe organ failure, on the list or already undergoing liver transplantation and referred for a dietetic visit.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
eating disorder | at the time of enrollment
  prevalence of eating disorders measured through validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Brodosi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Sant'Orsola, Bologna, BO, Italy